CLINICAL TRIAL: NCT01839617
Title: Early Versus Late Parenteral Nutrition in Cancer Patients Undergoing Abdominal Surgery
Brief Title: Study Comparing Early and Late Nutrition in Cancer Patients Undergoing Abdominal Surgery
Acronym: PaNCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Patrícia Camargo Marques, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICESP
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Cancer; Abdominal Surgery; Parenteral Nutrition
Keywords: parenteral nutrition; early nutrition; abdominal surgery; cancer
MeSH Terms: conditions — Neoplasms; Hyperphagia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (2):
- Early parenteral nutrition (Active Comparator): Parenteral nutrition starts at 2nd postoperative day.
  Interventions: Dietary Supplement: Early parenteral nutrition
- Late parenteral nutrition (Active Comparator): Parenteral nutrition starts at 7th postoperative day.
  Interventions: Dietary Supplement: Late parenteral nutrition

INTERVENTIONS:
Dietary Supplement: Early parenteral nutrition
  Arms: Early parenteral nutrition
Dietary Supplement: Late parenteral nutrition
  Arms: Late parenteral nutrition

SUMMARY:
The aim of this study is to find which is the best nutritional strategy in cancer patients undergoing abdominal surgery regarding postoperative complications.

DETAILED DESCRIPTION:
There is a controversy regarding the timing of initiation of parenteral nutrition in cancer patients undergoing abdominal surgery in whom caloric targets cannot be met by enteral nutrition alone.

This is a randomized and controlled trial comparing early initiation with late initiation of parenteral nutrition.

Early-initiation group: patients will be randomized to initiate parenteral nutrition in the 2nd day after surgery.

Late-initiation group: patients will be randomized to initiate parenteral nutrition in the 7th day after surgery.

Calculations regarding the caloric goal included protein energy and were based on corrected ideal body weight, age and sex. When oral or enteral nutrition covered 80% of the calculated caloric goal, parenteral nutrition was reduced and progressively stopped.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Laparotomy for abdominal cancer surgery: urological, gynecological, digestive, abdominal sarcomas and melanomas, lymphomas and abdominal vascular.
* Informed consent form signed by the patient or legal guardian.

Exclusion Criteria:

* Reoperation within one year from the previous surgery. using previously parenteral nutrition.
* Participation in another research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2018-04-10 (Estimated)

PRIMARY OUTCOMES:
Clinical complications | 30 days
  respiratory, cardiovascular, renal, neurological, infectious, surgical

SECONDARY OUTCOMES:
Mortality | 30 days
  30-day mortality
Length of stay in ICU and in hospital | 30 days
  Length of stay
ICU readmission rate | 30 days
  ICU readmission rate
Duration of pharmacologic hemodynamic support | 30 days
  duration of vasopressor therapy
Levels of C-reactive protein | 7 days
  serum levels of C-reactive protein
Duration of mechanical ventilation | 30 days
  Duration of invasive mechanical ventilation
Liver dysfunction | 30 days
  liver dysfunction according SOFA

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Marques, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (2):
- Brazil (2):
  - Cancer Institute of the State of Sao Paulo, São Paulo, São Paulo
  - ICESP, São Paulo, São Paulo